CLINICAL TRIAL: NCT05417204
Title: Role of Abdominothoracic Muscular Activity on Symptoms of Functional Dyspepsia
Brief Title: Abdominothoracic Muscular Tone in Functional Dyspepsia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: PR(AG)163/2022
Record Dates: First submitted 2022-06-08; First posted 2022-06-14 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Dyspepsia
Keywords: Functional dyspepsia; Abdominal distension
MeSH Terms: conditions — Dyspepsia

STUDY DESIGN:
Intervention Model Description: Adaptive design: a sample size calculation based on the primary outcome will be performed after 30 patients complete the post-intervention evaluation.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Correction of abnormal somatic response to a meal (Experimental): Biofeedback in patients with functional dyspepsia and abnormal somatic response to a probe meal
  Interventions: Behavioral: Abdominothoracic biofeedback
- Sham intervention in patients with normal somatic response to a meal (Active Comparator): Biofeedback in patients with functional dyspepsia and normal somatic response to a probe meal
  Interventions: Behavioral: Abdominothoracic biofeedback

INTERVENTIONS:
Behavioral: Abdominothoracic biofeedback — A standard biofeedback technique (3 sessions over a 4-week period) directed at controlling the muscular activity (postural tone) of the abdominal walls, will serve as active intervention in the experimental group, and as a sham intervention in the active comparator group.

SUMMARY:
Background. Patients with functional dyspepsia report symptoms after eating without detectable cause. A recent proof-of-concept study demonstrated that in healthy subjects, the activity of the abdominal walls influences perception of digestive sensations, specifically, intentional abdominal distension (by a maneuver of diaphragmatic contraction) increased bloating sensation in response to a probe meal.

Aim. To determine the role of the abdominothoracic muscular activity on symptoms of functional dyspepsia.

Design. Parallel study in dyspeptic patients who have an abnormal somatic response to a probe meal (experimental group), and patients who do not (control group), comparing the effect of abdominophrenic biofeedback on dyspeptic symptoms. The probe meal will consist in stepwise ingestion of a comfort meal (hot ham and cheese sandwich plus orange juice) up to maximal satiation.

Intervention. A standard biofeedback technique (3 sessions over a 4-week period) directed at controlling the muscular activity (postural tone) of the abdominal walls, will serve as active intervention in the experimental group, and as a sham intervention in the control (active comparator) group.

The study outcomes will be measured before, immediately after and at 6 months after biofeedback: 1) Clinical symptoms measured by scales during 7 consecutive days. 2) Responses to the probe meal: (a) sensations measured by scales; (b) changes in girth by adaptive belts; (c) diaphragmatic position by abdominal ultrasound.

Relevance. The identification of a pathophysiological mechanism of dyspeptic symptoms could serve as an objective marker for diagnosis and as a target for the development of mechanistic treatments.

ELIGIBILITY:
Inclusion Criteria:

* Rome IV Criteria for functional dyspepsia

Exclusion Criteria:

* organic gastrointestinal diseases
* obesity
* history of anosmia and ageusia
* alcohol abuse
* eating disorders

Age- and-sex-matched healthy subjects will be included in parallel to the 30 first patients, to determine the normal values of the response to the probe meal. Healthy subjects will not undergo the intervention.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Postprandial fullness | 7 days
  Change in postprandial fullness (measured on daily postprandial fullness scales graded from 0, i.e., not at all, to 10, i.e., extremely severe) during 7 consecutive days before and immediately after intervention.

SECONDARY OUTCOMES:
Tolerance of a probe meal | 60 minutes
  Change in the amount of a probe meal tolerated (Kcal consumed) before and after intervention.
Digestive well-being after a probe meal | 60 minutes
  Change in digestive well-being after a probe meal (measured on a scale graded from -5, i.e., extremely negative, to +5, i.e., extremely positive) before and after intervention
Postprandial fullness after a probe meal | 60 minutes
  Change in postprandial fullness after a probe meal (measured on a scale graded from 0, i.e., not at all, to 10, i.e., extremely severe) before and after intervention
Abdominal distension in response to a probe meal | 60 minutes
  Changes in the girth response to a probe meal (measured by adaptive belts) before and after intervention.
Diaphragmatic response to a probe meal | 60 minutes
  Changes in the diaphragmatic response to a probe meal (measured by ultrasound) before and after intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Livovsky DM, Barber C, Barba E, Accarino A, Azpiroz F. Abdominothoracic Postural Tone Influences the Sensations Induced by Meal Ingestion. Nutrients. 2021 Feb 18;13(2):658. doi: 10.3390/nu13020658. PMID 33670508